CLINICAL TRIAL: NCT05817292
Title: Characterization of the Vaginal Microbiota in Fertile Age: Correlations Clinical and Pathogenetic Correlations Among Gynecological Disorders.
Brief Title: Study of the Vaginal Microbiota in Women Under Fertile Age
Acronym: vaginalbiota
Status: Completed | Type: Observational
Sponsor: Universita degli Studi di Catania (Other)
Collaborators: ProBioEtna (Unknown)
Responsible Party: Principal Investigator, Agnese Maria Chiara Rapisarda, doctor, Universita degli Studi di Catania
Other Study IDs: 16/2022/PO
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Vaginal Disease
MeSH Terms: conditions — Vaginal Diseases | interventions — Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — vaginal discharge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Probiotic: Assumption of commercially available supplements containing probiotics
  Interventions: Dietary Supplement: Probiotics
- Control: No assumption of supplements containing probiotics
  Interventions: Other: No intervention

INTERVENTIONS:
Dietary Supplement: Probiotics — Assumption of commercial probiotics
  Groups: Probiotic
Other: No intervention — No assumption of probiotics
  Groups: Control

SUMMARY:
Characterization of the vaginal microbiota of women under fertile age and study of correlations with gynecological disorders

DETAILED DESCRIPTION:
The study aimed to characterize, in women under fertile age, the composition and dynamics of the vaginal microbiota as well as to in-depth study correlations among microbiota and gynecological disorders

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years;
* Presence of at least one vaginal sign or symptom (leucorrhoea, burning, itching, and subjective vaginal discomfort);
* Presence of at least 3 Amsel criteria;
* Nugent score ≥ 7;
* lactobacillary grade ≥ 2 (LBG) (according to Donders classification);
* presence of blastospores and/or pseudohyphae evaluated by fresh mount microscopy

Exclusion Criteria:

* Age < 18 years;
* Nugent score < 7;
* presence of sexually transmitted disease due to Chlamydia, Neisseria gonorrhoeae, or Trichomonas vaginalis as well as specific cervico-vaginitis or severe vulvovaginal symptoms related to acute candidiasis;
* Clinically apparent herpes simplex infection;
* Human papillomavirus or human immunodeficiency virus infections;
* Use of antibiotic, antifungal, probiotic, or immunosuppressive drugs during the past four weeks;
* Use of vaginal contraceptives;
* Pregnancy or breastfeeding, chronic diseases, neoplastic disease, diabetes, genital tract bleeding)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in fertile age
Study Population: healthy volunteers with vaginal microbiota imbalance
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Microbiota | Baseline; end of the treatment (10 days) ; wash-out (4 weeks)
  Change from baseline in the composition of the vaginal microbiota with the increase of the cell density of lactobacilli (at least 3 log units) and decrease of pathogens (at least 2 log units) at the end of the treatment (10 days) and during the wash-out period (4 weeks after the end of the treatment)
Signs | Baseline; end of the treatment (10 days) ; wash-out (4 weeks)
  Change from baseline of Amsel's criteria at the end of the treatment (10 days) and during the wash-out period (4 weeks after the end of the treatment)
Signs | Baseline; end of the treatment (10 days) ; wash-out (4 weeks)
  Change from baseline of the Nugent score with values between 0 and 3 at the end of the treatment (10 days) and during the wash-out period (4 weeks after the end of the treatment)
Symptomatology | Baseline; end of the treatment (10 days) ; wash-out (4 weeks)
  Change from baseline of vulvovaginal erythema/edema, vulvar discomfort, burning, and itching

SECONDARY OUTCOMES:
Wellbeing | Baseline; end of the treatment (10 days) ; wash-out (4 weeks)
  Change from baseline of the quality of life based on the Short Form-36 (SF-36) questionnaire. Values ranging from 0 to 100 indicate worst and better outcomes, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cianci, Prof, Study Director — University of Catania
Locations (1):
- University of Catania, Catania, Italy